CLINICAL TRIAL: NCT02105129
Title: A Phase I, Randomized, Double Blind, Placebo-controlled, Dose-escalating Study of the Safety, Tolerability and Pharmacokinetics of Single and Repeat Doses of HMPL-523
Brief Title: A Study of the Safety, Tolerability and Pharmacokinetics of HMPL-523
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014-523-00AU1
Record Dates: First submitted 2014-03-19; First posted 2014-04-07 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HMPL-523 (Experimental): Single/Multiple Ascending Dose. oral administration, a single dose of 5, 20, 50, 100, 200 and 300 mg (Part A) and multiple dose of HMPL-523 at dose level based on result of Part A
  Interventions: Drug: HMPL-523
- Placebo (Placebo Comparator): Placebo: oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HMPL-523 — HMPL-523: Oral administration with a single dose of 5, 20, 50, 100, 200 and 300 mg in Part A, followed by multiple doses of selected strength in Part B Other Name: NA
  Other Names: HMPL-523 acetate
  Arms: HMPL-523
Drug: Placebo — Oral administration
  Other Names: HMPL-523 Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of a single dose of up to 800 mg in Part A (evaluated in planned steps of 5, 20, 50, 100, 200, 300 mg under fasted conditions, followed by 300, 400, 600 and 800 mg HMPL-523 under fed conditions of a standard meal, followed by multiple doses of 200, 300, 400 and 500 mg of HMPL-523 in Part B, in healthy male volunteers.

The secondary objective is to determine the pharmacokinetic profile of single (Part A) and multiple (Part B) oral doses of HMPL-523 in healthy male volunteers and to determine the preliminary effect of food (Part C）

DETAILED DESCRIPTION:
This is a Phase I study with 3 parts:

Part A: Double blind, randomized, placebo-controlled, dose-escalating, single dose study in healthy volunteers.

Part B: Double blind, randomized, placebo-controlled, dose-escalating, multiple dose study in healthy volunteers.

Part C: Open labeled, single dose, cross-over, preliminary food effect study in healthy volunteers.

Number of subjects:

Part A: 80 healthy volunteers (10 cohorts of 8 subjects) Part B: About 40 healthy volunteers (5 cohorts of 8 subjects) In Part B, the multiple doses are 200(Cohort B1), 300(Cohort B2), 400(Cohort B3), and 500 mg(Cohort B4) and 8 subjects will be enrolled in each cohort. At dose 200mg, additional cohort (Cohort B1a) with 8 subjects needs to be enrolled based on the clinical data (safety, tolerability, available PK data and clinical laboratory values). The decision is made jointly by the Principal Investigator and the sponsor. Within each cohort, 6 subjects will receive HMPL-523 and 2 subjects will receive placebo Part C: 6 healthy volunteers (1 cohort; all will receive HMPL-523 100 mg).

Treatments:

-Part A: Single Ascending Dose.Subjects will receive a single dose of up to 800 mg HMPL-523 or matching placebo during Day 1. The planned dose levels are: 5, 20, 50,100, 200, 300 mg under fasted conditions, followed by 300, 400, 600, 800 mg under fed conditions with a standard meal, according to the randomization schedule. Dose levels may be repeated, reduced or administered as a split dose if deemed appropriate by the Principal Investigator and Sponsor's medical Expert.

For Cohort 1 a sentinel group (1 HMPL-523 and 1 placebo) will be dosed at 5 mg HMPL-523, 24 hours prior to the planned dosing of the remaining six subjects. Dosing of the remaining six will be based on investigator judgment. The decision to dose escalate will be made jointly by the Principal Investigator and the sponsor based on the clinical data (safety, tolerability, available PK data and clinical laboratory values).

-Part B: Multiple Ascending Dose (MAD). Part B of the study has been designed to assess the effects of multiple ascending doses of HMPL-523 in healthy volunteers. The total daily doses and dosing regimen for Part B have been determined as 200, 300,400 and 500 mg based on the review of safety and PK data from Part A, made jointly by the Principal Investigator and the sponsor. The dose will be the same or less than one already administered to participants in Part A. Because dog has similar protein binding to humans, we will closely monitor the clinical safety and laboratory result when the AUC is getting to 2085 h*ng/mL, which is the NOAEL AUC in dogs. Further dose escalation will be based on clinical safety and discussion between the sponsor and the investigators.

Part C: Preliminary Food Effect Study. Part C of the study has been designed to preliminarily assess the effect of food on the pharmacokinetics of HMPL-523 in healthy volunteers. Subjects will first receive a single dose of HMPL-523 100mg under fasted conditions (Period 1) and then following a washout period of 7 days, will receive a single dose of HMPL-523 100mg after consuming a standard high fat breakfast (fed conditions) (Period 2). Part C may be conducted at any time, provided 100 mg has been deemed safe in Part A.

Safety data:

The following safety evaluations will be performed during the study: Adverse events, physical examination, clinical safety laboratory (hematology, clinical chemistry, urinalysis), body weight, oral temperature, triplicate blood pressure and heart rate , and ECG .

ELIGIBILITY:
Inclusion Criteria:

* Informed consent must be obtained in writing for all subjects before enrollment into the study
* Healthy male subjects aged 18 to 45years inclusive at the time of screening
* Body mass index ≥19.0 and ≤ 30.0 kg/m2
* No clinically significant abnormalities as determined by medical history and physical examination, especially with regard to the liver, bile and gastrointestinal systems
* No clinically significant laboratory values and urinalysis, as determined by the clinical Investigator.
* No clinically significant findings in ECG, blood pressure and heart rate, as determined by the clinical Investigator.
* Willing to comply with the contraceptive requirements of the study and must not donate sperm during the study or for 3 months afterwards. Subjects must agree to use a condom or to abstain from sexual intercourse throughout the trial and for 30 days afterwards.

Exclusion Criteria:

* Family history of premature Coronary Heart Disease
* Any condition requiring the regular use of any medication
* Exposure to prescription medications or to drugs known to interfere with metabolism of drugs within 30 days prior to Day 1
* Exposure to any other medication, including over-the counter medications, herbal remedies and vitamins 14 days prior to first dose
* Participation in another study with any investigational drug in the 30 days preceding Day 1 of the study
* Treatment in the previous 3 months with any drug known to have a well defined potential for toxicity to a major organ
* Current smoker of more than 10 cigarettes or equivalent / day prior to commencing the study and unable to completely stop smoking during the study
* Be in the exclusion period of any previous study with investigational drugs
* Symptoms of a clinically significant illness in the 3 months before the study
* Presence or sequelae of gastrointestinal, liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs
* Chronic constipation or diarrhea, irritable bowel syndrome, inflammatory bowel disease, Hemorrhoids or anal diseases with regular or recent presence of blood in feces
* History of significant allergic disease (e.g. Allergic to medications) and acute phase of allergic rhinitis in the previous 2 weeks before randomization or any food allergy
* Blood or plasma donation of more than 500 ml during the previous 30 Days before randomization and/or more than 50 ml in the 2 weeks prior to screening
* Known positive test for HIV
* Known positive test for hepatitis B or C, unless caused by immunization
* Current evidence of drug abuse or history of drug abuse within one year before randomization
* History of alcohol abuse or active alcoholism as defined in Appendix A Definition of alcohol abuse
* Mental condition rendering the subject incapable to understand the nature, scope, and possible consequences of the study
* Adults under guardianship and people with restriction of freedom by administrative or legal decisions
* Unlikely to comply with the clinical study protocol; e.g. uncooperative attitude, inability to return for follow-up visits, and improbability of completing the study
* Subject is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To assess number of participants with adverse events as a measure of safety and tolerability during dose escalating | 6 months

SECONDARY OUTCOMES:
To measure the plasma concentration of HMPL-523 in single and repeated doses | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lickliter, MD, Principal Investigator — Nucleus Network Ltd; Yan Wu, MD, Study Director — Hutchison Medipharma Limited
Locations (1):
- Nucleus Network Limited, Melbourne, Victoria, Australia